CLINICAL TRIAL: NCT02121002
Title: A Multi-Center, Double-Blind, Vehicle-Controlled, Parallel-Group Study Comparing a Generic Diclofenac Sodium Topical Gel, 1% to Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% in the Treatment of Subjects With Osteoarthritis of the Knee
Brief Title: Study Comparing a Generic Diclofenac Sodium Topical Gel, 1% to Voltaren in the Treatment of Subjects With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amneal Pharmaceuticals, LLC (Industry)
Collaborators: Sristek Clinical Research Solutions Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-DCG-001
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2021-06-16 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-05

CONDITIONS: Osteoarthritis
Keywords: Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diclofenac Sodium Topical Gel, 1% (Experimental): Diclofenac Sodium Topical Gel, 1%. 4 gm, 4 times a day for 4 weeks
  Interventions: Drug: Diclofenac Sodium Topical Gel, 1%
- Voltaren Topical Gel, 1% (Active Comparator): Voltaren Topical Gel, 1%. 4 gm, 4 times a day for 4 weeks
  Interventions: Drug: Voltaren Topical Gel, 1%
- Vehicle Diclofenac Sodium Topical Gel (Placebo Comparator): Vehicle Diclofenac Sodium Topical Gel. 4 gm, 4 times a day for 4 weeks
  Interventions: Drug: Vehicle Diclofenac Sodium Topical Gel

INTERVENTIONS:
Drug: Diclofenac Sodium Topical Gel, 1% — Opaque, white gel
  Arms: Diclofenac Sodium Topical Gel, 1%
Drug: Voltaren Topical Gel, 1% — Opaque, white gel
  Arms: Voltaren Topical Gel, 1%
Drug: Vehicle Diclofenac Sodium Topical Gel — Opaque, white gel
  Arms: Vehicle Diclofenac Sodium Topical Gel

SUMMARY:
To establish the therapeutic equivalence and safety of a generic Diclofenac Sodium Topical Gel, 1% with Voltaren® Gel 1% in subjects with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, ambulatory male or non-pregnant female subjects aged ≥ 35 years with a clinical diagnosis of OA of the knee.
* Had an X-ray of the target knee, taken no more than 1 year before baseline, showing evidence of OA with Kellgren-Lawrence grade 1-3 disease.
* After discontinuing all pain medications for at least 7 days, has at least moderate pain on movement for target knee
* If female and of child-bearing potential, agree to abstain from sexual intercourse or use a reliable method of contraception during the study
* Able to tolerate rescue medication with paracetamol/acetaminophen.

Exclusion Criteria:

* Pregnant or lactating or planning to become pregnant during the study period.
* X-ray showing evidence of OA with Kellgren-Lawrence grade 4 disease.
* History of OA pain in the contralateral knee requiring medication within 1 year prior to screening.
* After discontinuing all pain medications for at least 7 days, has a baseline score of ≥20 mm on a 0-100 mm Visual Analog Scale (VAS) for the contralateral knee immediately prior to randomization.
* History of secondary OA, rheumatoid arthritis, chronic inflammatory disease or fibromyalgia.
* History of asthma, hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function or liver disease.
* History of gastrointestinal bleeding or peptic ulcer disease.
* Use of warfarin or other anticoagulant therapy within 30 days of study randomization.
* Elevated transaminases at screening.
* Use of ACE inhibitors, cyclosporine, diuretics, lithium or methotrexate, within 30 days of study randomization.
* Concomitant use of corticosteroids or use within 30 days of study randomization.
* Concomitant acetylsalicylic acid therapy other than a stable low dose used for cardiac prophylaxis taken for at least 3 months prior to enrollment and maintained throughout the duration of the study.
* Known allergy to aspirin or nonsteroidal anti-inflammatory drug
* Any other acute or chronic illness that could compromise the integrity of study data or place the subject at risk by participating in the study.
* Receipt of any drug as part of a research study within 30 days prior to screening.
* Previous participation in this study.
* Any use between screening and baseline of a treatment or medication that may potentially confound study assessment that may potentially confound study assessment (e.g. use of topical analgesics or anti-inflammatory drugs).
* Recent history of major knee injury or surgery.
* Known history of positive HIV

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1176 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prayag Shah, MD, Study Director — Amneal Pharmaceuticals, LLC
Locations (22):
- India (22):
  - Sunshine Hospitals, Secunderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Rathi Orthopedic and Research Centre, Ahmedabad, Gujarat
  - B. J. Medical College & Hospital, Ahmedabad, Gujarat
  - GMERS Medical College and Hospital, Ahmedabad, Gujarat
  - Shir Hatkesh Sarvajanik Tabibi Chikitsha Kendra, Jūnāgadh, Gujarat
  - Centre For Knee Surgery, Vadodara, Gujarat
  - Shree Giriraj Multispeciality Hospital, Rajkot, Gujurat
  - St Johns Medical College, Bangalore, Karnataka
  - K L E Societys Jawaharlal Nehry Medical College, Belagavi, Karnataka
  - Mysore Medical College, Mysore, Karnataka
  - Government Medical College, Calicut, Calicut, Kerala
  - Psm Dept Ltmmc & Ltmg Hospital, Mumbai, Maharashtra
  - Government Medical College, Nagpur, Maharashtra
  - Jasleen Hospital, Nagpur, Maharashtra
  - Lata Mangeshkar Hospital, Nagpur, Maharashtra
  - Bj Medical College, Pune, Maharashtra
  - Malpani Multispeciality Hospital, Jaipur, Rajasthan
  - Apollo Speciality Hospitals, Madurai, Tamil Nadu
  - M V Hospital and Research Centre, Lucknow, Uttar Pradesh
  - King Georges Medical University, Lucknow, Uttar Pradesh
  - Goa Medical College, Goa

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Diclofenac Sodium Topical Gel, 1% | Voltaren Topical Gel, 1% | Vehicle Diclofenac Sodium Topical Gel
Started | 392 | 393 | 391
Completed | 385 | 389 | 381
Not Completed | 7 | 4 | 10
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 4
Not completed — Protocol Violation | 1 | 2 | 4
Not completed — Concomitant therapy | 0 | 1 | 1
Not completed — Others | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline participants in the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Diclofenac Sodium Topical Gel, 1% | Voltaren Topical Gel, 1% | Vehicle Diclofenac Sodium Topical Gel | Total
Number analyzed (Participants) | 391 | 393 | 391 | 1175
Age, Customized [Number; unit: Participants]
  <= 18 years | 0 | 0 | 0 | 0
  between 18 and 65 years | 357 | 351 | 354 | 1062
  >=65year | 34 | 42 | 37 | 113
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 255 | 244 | 254 | 753
  Male | 136 | 149 | 137 | 422

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 4 Weeks in WOMAC Pain Score
Description: Mean change from baseline to week 4 in the Western Ontario McMaster
  Osteoarthritis (WOMAC) pain score:
  5-point Likert scale: none=o, mild=1, moderate=2, severe=3, extreme=4
Time Frame: Baseline and Week 4
Population: Across study groups, the per protocol (PP) population included 1147 subjects (97.53%) and the modified intention-to-treat (mITT) population included 1166 subjects (99.15%).
  For various reasons, 10 subjects were excluded from mITT population while 29 subjects were excluded from PP population out of 1176 subjects randomized in the study
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Diclofenac Sodium Topical Gel, 1% | Voltaren Topical Gel, 1% | Vehicle Diclofenac Sodium Topical Gel
Number analyzed (Participants) | 391 | 393 | 391
score on a scale | 2.2332 (0.1160) | 2.0287 (0.1157) | -0.6387 (0.1172)

ADVERSE EVENTS:
Time Frame: The over all time frame for any the Adverse Events is maximum 9days starting from date of appearance to date of disappearance.
Arm/Group | Diclofenac Sodium Topical Gel, 1% | Voltaren Topical Gel, 1% | Vehicle Diclofenac Sodium Topical Gel
All-Cause Mortality (participants affected / at risk) | 0/391 | 0/393 | 0/391
Serious Adverse Events (participants affected / at risk) | 0/391 | 0/393 | 0/391
Other Adverse Events (participants affected / at risk) | 2/391 | 2/393 | 3/391
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diclofenac Sodium Topical Gel, 1% (N=391) | Voltaren Topical Gel, 1% (N=393) | Vehicle Diclofenac Sodium Topical Gel (N=391)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema, (General disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis Cough (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus and Rash Pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No